CLINICAL TRIAL: NCT01714271
Title: Promotora-based Latino Family CVD Risk Reduction: Remaking the Home Environment
Brief Title: Promotora-based Latino Family CVD Risk Reduction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Southern California (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1P50HL105188-6094; 1P50HL105188 (NIH)
Record Dates: First submitted 2012-10-20; First posted 2012-10-25 (Estimated); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Heart Disease; Cancer
MeSH Terms: conditions — Heart Diseases; Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home environs-based lifestyle counseling (Experimental): Home environs-based lifestyle counseling Involves Spanish-speaking community health workers interacting with intervention subjects in home visits and phone calls - 12 contacts overall. The counseling focuses on promoting subject adherence to the Dietary Guidelines for Americans (DGA) and the Physical Activity Guidelines for Americans (PAGA) with special attention devoted to changing the home environment to make it optimally supportive of the lifestyle choices consistent with the DGA and PAGA. Study participants will also be provided 4 group education sessions that will be devoted to improving subject adherence to the DGA and PAGA.
  Interventions: Behavioral: Home environs-based lifestyle counseling
- Cancer early detection (Experimental): Cancer Early Detection Spanish-speaking health educators will interact with study participants via a home visit and four telephone calls. The focus of the health education will be on practical strategies to detect cancer early to help prevent death from cancer. Cancer sites of interest will be: breast, cervical, skin, colon, prostate and testicular cancers. In addition, study participants will be provided two group education classes that will focus on the basics of the cancer process and why early detection and intervention can be life-saving.
  Interventions: Behavioral: Cancer early detection

INTERVENTIONS:
Behavioral: Home environs-based lifestyle counseling — Social learning theory-based behavior modification embedded in a social ecological framework is used to shape both the home environment and the lifestyle choices of the study participants to optimize their adherence to the Dietary Guidelines for Americans and the Physical Activity Guidelines for Americans.
  Arms: Home environs-based lifestyle counseling
Behavioral: Cancer early detection — Conventional health education is used to increase study participant knowledge of practical strategies for detecting and treating common cancers early, before cancers have metastasized. Additional instruction is devoted to the biology and physiology of the cancer process. Although some mention will be made of the importance of maintaining a healthy weight for minimizing lifetime risk of certain cancers, most of the focus will be on episodic cancer screening, e.g., mammograms, PAP smears, colonoscopies, etc. for prevention of death from cancer.
  Arms: Cancer early detection

SUMMARY:
This family environment-focused health behavior change intervention is being carried out by extensively trained community health workers (promotores) familiar with the community in East Los Angeles. The hypothesis being tested is that home environment-focused health behavior change will reduce risk of arterial stiffness, an early-in-life predictor of heart disease. The community health workers will provide most of the health promotion counseling. The promotores will provide up to 16 counseling sessions to a designated adult family member without diabetes. The sessions will focus on improving the home environment in order to reduce television viewing, increase fruit and vegetable intake, decrease intake of refined carbohydrates, prompt more frequent monitoring of body weight and increase daily physical activity. The lifestyle change goals will be tailored to the families' capacity for change and will be consistent with the Dietary Guidelines for Americans, especially the MyPlate.gov messages, the Dietary Approaches to Stop Hypertension (DASH) diet and at least 30 minutes of daily moderate physical activity.

DETAILED DESCRIPTION:
This is a randomized controlled trial involving non-diabetic residents of East Los Angeles, most of whom are low-income, mostly immigrant Mexican Americans. The family environment-focused health behavior change intervention is being carried out by extensively trained community health workers (promotores) familiar with the community in East Los Angeles. The comparison condition is a more traditional health education approach to teaching residents about practical early cancer detection strategies designed to reduce risk of death from cancer.

The hypothesis being tested is that home environment-focused health behavior change will reduce risk of arterial stiffness, an early-in-life predictor of heart disease. The community health workers will provide most of the health promotion counseling. The promotores will provide up to 16 counseling sessions to a designated adult family member without diabetes. The sessions will focus on improving the home environment in order to reduce television viewing, increase fruit and vegetable intake, decrease intake of refined carbohydrates, prompt more frequent monitoring of body weight and increase daily physical activity. The lifestyle change goals will be tailored to the families' capacity for change and will be consistent with the Dietary Guidelines for Americans, especially the MyPlate.gov messages, the Dietary Approaches to Stop Hypertension (DASH) diet and at least 30 minutes of daily moderate physical activity.

Secondary outcomes include: aerobic fitness, fruit and vegetable intake as assessed by food frequency questionnaire, endothelial function, body mass index, waist circumference, blood pressure, a metabolic syndrome score, and quality of life. Relative to the cancer early detection condition, the lifestyle change intervention is expected to improve fitness, increase fruit and vegetable intake, improve endothelial function, improve BMI, reduce excess waist circumference, improve blood pressure, and improve quality of life.

If results confirm hypotheses, the results will support investing more public health resources into environmental and policy strategies design to make it easier for populations to adhere to the Dietary Guidelines for Americans and the Physical Activity Guidelines for Americans.

ELIGIBILITY:
Inclusion Criteria:

* Resides in East Los Angeles
* Home includes family member (spouse or 1st degree relative)who has been diagnosed with type 2 diabetes

Exclusion Criteria:

* BMI>40;
* Any condition that prevents engaging in daily physical activity / walking;
* pregnant;
* breast feeding;
* cardiovascular (CVD) event within 12 months;
* cancer requiring chemotherapy;
* other medical condition requiring active lifestyle intervention/dialysis;
* severe CVD or other disease known to significantly limit life expectancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2010-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in arterial stiffness as measured by pulse wave velocity | baseline, 6, 12, 24 months follow-up
  Pulse wave velocity is a measure of arterial stiffness that is sensitive to changes in health-related lifestyle changes.
Change in arterial stiffness as measured by the Augmentation index | baseline, 6, 12 and 24 months follow-up
  Augmentation index is another measure of arterial stiffness, also sensitive to changes in health-related lifestyle behaviors.

SECONDARY OUTCOMES:
Change in fasting glucose | baseline, 6, 12, 24 months
  Fasting blood glucose
Changes in glycosylated hemoglobin A1c (HbA1c) | baseline, 6, 12, 24 months follow-up
  Glycosylated hemoglobin A1c. Measure of glucose control over several months.
Changes in answers to MyPlate evaluation questions | baseline, 6, 12, 24 months follow-up
  Self-report questions about adherence to MyPlate.gov recommendations. These include questions about daily fruit intake, vegetable intake, replacement of sugary beverages with water, effort to make at least 1/2 of grain intake whole grain, effort to seek out lower sodium options, and daily intake of non-fat or low-fat milk.
Changes in food frequency measure of fruit and vegetable intake | Baseline, 6, 12, 24 months follow-up
  Block Food Frequency assessment conducted in Spanish by interview. Information will include estimate of total fruit and vegetable intake over the last 6 months.
Changes in waist circumference | baseline, 6, 12 and 24 months
  Measure of waist circumference, a common predictor of cardiovascular risk
Change in aerobic capacity | Baseline, 6, 12, 24 months
  Bruce protocol treadmill test. Estimate the VO2max (maximum aerobic capacity) using Foster's equation.
Change in metabolic syndrome score | Baseline, 6, 12, 24 months
  Metabolic syndrome marker levels. The ATP III criteria for metabolic syndrome markers include:
  * sex-specific excess waist circumference (men > 102 cm, women >88 cm),
  * fasting plasma triglycerides >= 120 mg/dl,
  * fasting plasma HDL(men)<40 or (women)<50 mg/dl,
  * blood pressure >=135/85,
  * fasting glucose >=110 mg/dl). Each subject's metabolic syndrome marker level can range between zero and five, with zero representing no metabolic syndrome risk and five representing maximum risk. The a priori expectation is that each marker will be treated as equally important but this study will provide the opportunity to examine this assumption critically.
Change in plasma lipids | Baseline, 6, 12, 24 months
  Plasma lipids to be measured include LDL-cholesterol, HDL-cholesterol and triglycerides. Blood samples will be obtained by venipuncture.
Change in blood pressure | Baseline, 6, 12, 24 months
  Blood pressure will be assessed in study participants sitting quietly by trained personnel using regularly calibrated sphygmomanometry.
Change in physical activity assessment | Baseline, 6, 12, 24 months
  International Physical Activity Questionnaire - short form (IPAQ-short). Questions ask about the number of days in the last 7 days that the participant exercised vigorously or moderately vigorously. Follow-up questions query the participant about the time (minutes & hours) spent per day in doing vigorous or moderately vigorous physical activity on those days when they exercised.
Change in body mass index (BMI) | Baseline, 6, 12, 24 months
  Body mass index (BMI) obtained by taking the ratio of measured weight (kg) to measured height (m). Weight is obtained using a regularly calibrated balance beam scale. Height is obtained using a stationary stadiometer.
Change in quality of life | Baseline, 6, 12, 24
  The SF-12 is a well-accepted short form of the well-known SF-36 quality of life instrument.
Change in weight loss strategies | Baseline, 6, 12, 24
  Questionnaire includes 11 items that query the participant about weight control strategies used in the last year, including: exercise, restricting calories, fasting, diet pills, vomiting / laxative use, joining a gym, joining a commercial weight loss program such as WeightWatchers, meal replacement products, herbal medicines, diet bars, restriction on TV watching.
Change in endothelial function | Baseline, 6, 12, 24 months
  Flow-mediated dilation is the most widely used non-invasive test for assessing endothelial function, that is, the functional status of the inner lining of the major blood vessels. This technique measures endothelial function by inducing reactive hyperemia (blood volume expansion) via temporary arterial occlusion (blocking blood flow with inflated blood pressure cuff) and measuring the resultant relative increase in blood vessel diameter via ultrasound.
Change in self-efficacy to adhere to DASH-style dietary pattern | Baseline, 6, 12, 24 months
  List of 10 self-efficacy items that assess the study participant's confidence that she/he can adhere to various features of the Dietary Approaches to Stop Hypertension (DASH) diet.
Change in mental health status | Baseline, 6, 12, 24
  Mental health index-5 (MHI-5) consists of 5 questionnaire items designed to assess emotional well-being.

CONTACTS AND LOCATIONS:
Overall Officials: William J McCarthy, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Roybal Comprehensive Health Center, Los Angeles, California, United States